CLINICAL TRIAL: NCT06599983
Title: Educational Storytelling, an Innovative Interdisciplinary Program Against Child Maltreatment
Acronym: EST program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oral Health Centre of Expertise in Western Norway (Other)
Collaborators: Educational storytelling forlag og film (Unknown)
Responsible Party: Principal Investigator, Ingfrid Vaksdal Brattabø, PhD researcher, Oral Health Centre of Expertise in Western Norway
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Educational Storytelling
Record Dates: First submitted 2024-03-15; First posted 2024-09-19 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Child Abuse; Child Neglect; Child Sexual Abuse; Child Maltreatment; Oral Health; Dental Neglect
Keywords: Educational program; Child abuse and neglect; Detection; Reporting; Knowledge; Prevention; Evaluation; Dental professionals; Child welfare services; Child protection

STUDY DESIGN:
Intervention Model Description: The aim of this study, is to evaluate if the novel educational program for dental personnel: Educational Storytelling, an Educational Program Against Child Abuse and Neglect has any effect. A total of 39 public dental health clinics in Vestland county Norway, were randomized into two groups, test and control groups.
  The dental clinics in the test group attended the program, Educational Storytelling, an Educational Program Against Child Abuse and Neglect. The control grup did not attend any program.
  Both test and control group recieved a total of 3 questionnaires by e-mail in the following timeframe:
  * Three weeks before the test group attended the educational program.
  * One week after the test group attended the educational program
  * Six months after the test group attended the educational program.
  A few months after the last questionnaire was closed, the dental clinics allocated in the control group, attended the educational program
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test group (Experimental): The test group attended the one day educational programme, Educational Storytelling, an Educational Program Against Child Abuse and Neglect.
  Interventions: Other: Educational program, Educational Storytelling, an Educational Program Against Child Abuse and Neglect.
- Control group (No Intervention): The control group did not attend the one day educational programme, Educational Storytelling, an Educational Program Against Child Abuse and Neglect.

INTERVENTIONS:
Other: Educational program, Educational Storytelling, an Educational Program Against Child Abuse and Neglect. — One day educational program, aiming at increase dental personnels attitude, knowledge and behaviour in regard to detect and report child abuse and neglect, and to treat patients with known and unknown history of child abuse and neglect.
  Arms: Test group

SUMMARY:
Educational Storytelling, an Innovative Novel Interdisciplinary Program Against Child Maltreatment, is developed for dental personnel. The program aims at increasing dental personnels ability to detect, report and treat patients being victims of child abuse or neglect.

The objectives of the program is to contribute to the fulfillment of the Norwegian:

* Dental health services act

  §1-3 c The dental health service responsibility to prevent, detect and avert violence and sexual abuse
* Health Personnel act §33 Obligation to report suspected cases of child maltreatment to child welfare services.

The Educational Storytelling program aims to increase the dental health personnels knowledge and competence related to:

* Detecting child abuse and neglect.
* Reporting suspected cases of child maltreatment to child welfare services.
* Treatment of patients with known and unknown history of child abuse and neglect, trauma sensitive dental treatment.

The aim of this trial is to evaluate if the educational program has any effect.

DETAILED DESCRIPTION:
Educational Storytelling, an Innovative Novel Interdisciplinary Program Against Child Maltreatment, is a blended mode learning tool. The program combines a digital platform including documentary film, expert interviews and research findings with on site teaching, group work, reflections and discussions delivered by moderators. The program has a collective focus, contributing to the development of a shared understanding and social norm at the workplace.

The digital program consists of 7 chapters which covers different topics.

1. Introduction.
2. Documentary film, All that I am.
3. The dental health personnels role in detection of child abuse, and neglect.
4. Trauma sensitive treatment.
5. Learn more about trauma.
6. Childrens advocacy center and ethical platform for professionals.
7. Wrapping up.

The chapters include interview with different experts, group work, reflection tasks, research findings and supplementary material.

Each program participant gets an unique access to the digital program for two years.

The programs estimated completion time, including lunch is 7,5 hours. The program gives 6 continuing education credits from the Norwegian dental association (Norsk tannlegeforening) .

The educational program has been developed based on research findings from the public dental health service in Norway, in regard to their experience with detection of child abuse and neglect, reporting to and collaborating with child welfare services.

In order to measure if the program has any effect, a cluster randomized controlled trial has been conducted.

ELIGIBILITY:
Inclusion Criteria:

Working in the public dental health service in Vestland county

-

Exclusion Criteria:

Not working in the public dental health service in Vestland county

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 430 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Questionnaire, assessing attitude, knowledge and behaviour among dental health personnel in regard to talk to children that one suspect is being a victim of child abuse and neglect | Two weeks pre, one week and 6 months after program attendance
  To assess dental health personnels attitude, knowledge and behaviour in regard to talk to children that one suspect is being a victim of child abuse and neglect different questions were used.
  Example:
  How unimportant/important is it for you to have a good understanding of how best to talk to children you suspect are victims of child abuse or neglect (to increase prospect of child confiding)?
  Response options: (7 point scale, (1) very unimportant to (7) very important)
  How unsure/ sure are you on how best to talk with children that you suspect are being victim of child abuse or neglect ( in order to increase prospect of child confiding) Response options:(7 point scale, (1)very unsure to (7)very sure )
Questionnaire, assessing behaviour among dental health personnel in regard to suspect and report casese of child abuse and neglect to child welfare services | Two weeks pre, 6 months post program attendance
  In order to assess reporting behaviour, questions focusing on dental personnels experience with:
  * suspecting child abuse and neglect.
  * reporting child abuse and neglect.
  * failing to report child abuse and neglect. during career, and previous 6 months were used.
  Example:
  In the past 6 months, have you sent a report of concern to child welfare services because you suspected that a child (aged 0-18) was suffering child abuse or neglect?
  Response options: Yes or No.
  If yes:
  Please state how many times you have sent a report of concern to child welfare services (in the past 6 months) when suspecting that a child (aged 0-18) was suffering child abuse or neglect.
Questionnaire, assessing attitude, knowledge and behaviour among dental health personnel in regard to provide trauma sensitive treatment | Two weeks pre, one week and 6 months after program attendance
  In order to assess attitude, knowledge and behaviour in regard to provide trauma sensitive treatment to children that one suspect is being a victim of child abuse and neglect different questions were used.
  Example:
  How unconfident /confident are you in your ability to identify whether a patient needs trauma-informed care? Response options:(7 point scale, (1)very unconfident to (7)very confident)
  How unsure/ sure are you in regard to provide trauma sensitive treatment? Response options:(7 point scale, (1)very unsure to (7)very sure )
  Over the course of an average month, roughly how many patients (aged 0-100) do you see who need trauma-informed care? Each patient should only be counted once regardless of how many appointments they attend.
  Response options: (3 point scale, (1)none, (2)=fewer one per month, (3) one or more patients per month.)
  If (3): Please enter roughly how many patients (aged 0-100) you see per month who need trauma-informed care.
Questionnaire, assessing dental health personnels attitude, social norm, perceived behaviour control and behaviour in regard to detect and report child abuse and neglect to child welfare services. | Two weeks pre, one week and 6 months post program attendance
  To assess dental health personnels attitude, social norm, perceived behaviour control and behaviour in regard to detect and report child abuse and neglect to child welfare services questions in line with The Reason Action Approach (RAA), by M. Fishbein and I. Ajzen (2010) were used. The questions assess dental health personnels experiental attitude, instrumental attitude, descriptive norm, injunctive norm, capacity, autonomy, intention and behaviour.
  Example:
  The following people would send a report of concern if they came to suspect child abuse or neglect over the next 6 months:
  * my colleagues at the clinic.
  * most people in my situation.
  If, over the next 6 months, I come to suspect child abuse or neglect, the following people would think that I should send a report of concern:
  * my colleagues at the clinic.
  * most people who matter to me.
  Response options: (7 point scale, (1) completely disagree to (7) completely agree)

CONTACTS AND LOCATIONS:
Overall Officials: Ingfrid V Brattabø, PhD, Principal Investigator — Oral Health Centre of Expertice Western Norway
Locations (1):
- Ingfrid Vaksdal Brattabø, Stanghelle, Norway

IPD SHARING:
Plan to Share IPD: No